CLINICAL TRIAL: NCT01533428
Title: A Phase III, Double-blind, Randomized, Placebo-controlled, Multicenter Study Evaluating the Efficacy and Safety of QUTENZA® in Subjects With Painful Diabetic Peripheral Neuropathy
Brief Title: A Study to Evaluate Efficacy and Safety of a Single Application of Capsaicin 8%Transdermal Delivery System Compared to Placebo in Reducing Pain Intensity in Subjects With Painful Diabetic Peripheral Neuropathy (PDPN)
Acronym: STEP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: E05-CL-3004
Record Dates: First submitted 2012-02-12; First posted 2012-02-15 (Estimated); Results first posted 2015-03-13 (Estimated); Last update posted 2015-11-04 (Estimated); Status verified 2015-10

CONDITIONS: Diabetic Peripheral Neuropathy; Pain
Keywords: Painful Diabetic Peripheral Neuropathy,; Capsaicin 8% transdermal delivery system
MeSH Terms: conditions — Pain | interventions — Capsaicin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Capsaicin 8% (Experimental): Capsaicin 8% patch was applied for 30 minutes to the painful area(s) on Day 1
  Interventions: Drug: Capsaicin 8%
- Placebo (Placebo Comparator): Placebo patch was applied for 30 minutes to the painful area(s) on Day 1
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Capsaicin 8% — Capsaicin 8% transdermal delivery system
  Other Names: Qutenza
  Arms: Capsaicin 8%
Drug: Placebo — Placebo Patch
  Arms: Placebo

SUMMARY:
The purpose of the study is to assess efficacy and safety of a single treatment of Capsaicin 8% transdermal delivery system in reducing pain from damaged nerves (neuropathic pain) caused by diabetes.

DETAILED DESCRIPTION:
Participants were divided into 2 groups of approximately equal size. In the first group, participants received a Capsaicin 8% patch applied for 30 minutes to the feet; in the second group, participants received a placebo patch applied for 30 minutes to the feet. Participants were involved in the study for approximately 12 weeks and have visited the clinic approximately 6 times.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of painful, distal, symmetrical, sensorimotor polyneuropathy which is due to diabetes, for at least 1 year prior to screening visit
* Average Numeric Pain Rating Scale (NPRS) score over the last 24 hours of ≥4 at the screening and the baseline visit

Exclusion Criteria:

* Primary pain associated with PDPN (Painful Diabetic Peripheral Neuropathy) in the ankles or above
* Pain that could not be clearly differentiated from, or conditions that might interfere with the assessment of PDPN (Painful Diabetic Peripheral Neuropathy), neurological disorders unrelated to diabetic neuropathy (e.g., phantom limb pain from amputation); skin condition in the area of the neuropathy that could alter sensation (e.g., plantar ulcer)
* Current or previous foot ulcer as determined by medical history and medical examination
* Any amputation of lower extremity
* Severe renal disease as defined by a creatinine clearance of <30 ml/min calculated according to the Cockcroft-Gault formula
* Clinically significant cardiovascular disease within 6 months prior to screening visit defined as cerebrovascular accident, unstable or poorly controlled hypertension, transient ischemic attack, myocardial infarction, unstable angina, current arrhythmia, any heart surgery including coronary artery bypass graft surgery, percutaneous coronary angioplasty/stent placement, or valvular heart disease
* Significant peripheral vascular disease (intermittent claudication or lack of pulsation of either the dorsalis pedis or posterior tibial artery, or ankle-brachial systolic blood pressure index of <0.80)
* Clinically significant foot deformities, including hallux rigidus, hallux valgus, or rigid toe as determined by physical examination as judged by the investigator
* Clinically significant ongoing, uncontrolled or untreated abnormalities in cardiac, renal, hepatic, or pulmonary function that may interfere either with the ability to complete the study or the evaluation of adverse events
* Diagnosis of any poorly controlled major psychiatric disorder
* Active substance abuse or history of chronic substance abuse within 1 year prior to screening visit or any prior chronic substance abuse (including alcoholism) likely to re-occur during the study period as judged by the investigator
* Hypersensitivity to capsaicin (i.e., chili peppers or over-the-counter [OTC] capsaicin products), any Capsaicin 8% transdermal delivery system excipients, Eutectic Mixture of Local Anaesthetics (EMLA) ingredients or adhesives
* Use of any topical pain medication, such as non-steroidal anti-inflammatory drugs, menthol, methyl salicylate, local anesthetics, steroids or capsaicin products on the painful areas within 7 days preceding the first patch application at the baseline visit
* Use of oral or transdermal opioids exceeding a total daily dose of morphine of 80 mg/day, or equivalent; or any parenteral opioids, regardless of dose, within 7 days preceding the first patch application at the baseline visit
* Skin areas to be treated with Capsaicin 8% transdermal delivery system showing changes such as crusting or ulcers
* Planned elective surgery during the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 369 (Actual)
Dates: Start 2012-02; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Study Manager, Study Chair — Astellas Pharma Europe B.V.
Locations (29):
- United States (29):
  - Site: 125, Anniston, Alabama
  - Site: 131, Fresno, California
  - Site: 123, Long Beach, California
  - Site: 116, Los Angeles, California
  - Site: 112, Orange, California
  - Site: 130, Walnut Creek, California
  - Site: 113, Milford, Connecticut
  - Site: 119, New London, Connecticut
  - Site: 117, Boynton Beach, Florida
  - Site: 124, Bradenton, Florida
  - Site: 107, Clearwater, Florida
  - Site: 120, Jupiter, Florida
  - Site: 108, Orlando, Florida
  - Site: 132, Oviedo, Florida
  - Site: 127, St. Petersburg, Florida
  - Site: 122, Tampa, Florida
  - Site: 133, Honolulu, Hawaii
  - Site: 126, New Bedford, Massachusetts
  - Site: 115, Ann Arbor, Michigan
  - Site: 128, Hazelwood, Missouri
  - Site:111, New York, New York
  - Site: 110, Winston-Salem, North Carolina
  - Site: 121, Kettering, Ohio
  - Site:106, Dallas, Texas
  - Site: 118, Houston, Texas
  - Site: 114, Houston, Texas
  - Site: 103, Lubbock, Texas
  - Site: 105, San Antonio, Texas
  - Site: 102, San Antonio, Texas

REFERENCES:
- [Derived] Simpson DM, Robinson-Papp J, Van J, Stoker M, Jacobs H, Snijder RJ, Schregardus DS, Long SK, Lambourg B, Katz N. Capsaicin 8% Patch in Painful Diabetic Peripheral Neuropathy: A Randomized, Double-Blind, Placebo-Controlled Study. J Pain. 2017 Jan;18(1):42-53. doi: 10.1016/j.jpain.2016.09.008. Epub 2016 Oct 13. PMID 27746370
- See also: Link to results on Astellas Clinical Study Results Web site — https://www.astellasclinicalstudyresults.com/study.aspx?ID=E05-CL-3004

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Capsaicin 8% | Placebo
Started | 186 | 183
Completed | 177 | 175
Not Completed | 9 | 8
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 2 | 1
Not completed — Withdrawal by Subject | 7 | 6

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set
Groups:
- Total: Total of all reporting groups
Arm/Group | Capsaicin 8% | Placebo | Total
Number analyzed (Participants) | 186 | 183 | 369
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.90 (10.64) | 62.00 (10.81) | 63.00 (10.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 82 | 154
  Male | 114 | 101 | 215
Race/Ethnicity, Customized [Number; unit: participants]
  White | 132 | 131 | 263
  Black or African American | 36 | 38 | 74
  Asian | 4 | 4 | 8
  American Indian or Alaskan Native | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 3
  Other | 11 | 7 | 18
Duration of Painful Diabetic Peripheral Neuropathy (PDPN) [Mean (Standard Deviation); unit: years] | 5.83 (4.01) | 5.72 (3.98) | 5.78 (3.99)
Glycosylated Hemoglobin (HbA1c) [Mean (Standard Deviation); unit: Percentage of Glycosylated Hemoglobin] | 7.39 (1.309) | 7.23 (1.223) | 7.31 (1.268)
Average Pain Score [Mean (Standard Deviation); unit: units on a scale] — Average pain was assessed by the Brief Pain Inventory-Diabetic Neuropathy (BPI-DN) on a numeric rating scale from 0 - 10, with 0 describing "no pain" and 10 describing severe pain listed as "pain as bad as you can imagine".
  units on a scale | 6.64 (1.416) | 6.38 (1.473) | 6.51 (1.449)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in the Average Daily Pain Score From Baseline to Between Weeks 2 and 8
Description: Percent change in the average daily pain score from baseline to between Weeks 2 and 8, measured using Question 5 of the Brief Pain Inventory-Diabetic Neuropathy (BPI-DN). Participants assessed their pain due to diabetes in the last 24 hours on a numeric rating scale from 0 (no pain) to 10 (pain as bad as you can imagine).
Time Frame: Baseline to between Weeks 2 to 8
Population: Intention to Treat (ITT); Baseline Last Observation Carried Forward (BLOCF) imputation was used.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Capsaicin 8% | Placebo
Number analyzed (Participants) | 186 | 183
percentage change | -27.44 (26.79) | -20.85 (28.92)
Statistical Analysis 1: Comparison: Capsaicin 8% vs Placebo; All statistical comparisons were made using two-sided tests at the 5% significance level; Test type: Superiority or Other; p = 0.025, ANCOVA; Analysis of covariance model including treatment, gender, pain score at baseline, HbA1c at screening and site as factors/covariates; LS Mean Difference = -6.6, 95% CI 2-sided [-12.3 to -0.8]

2. Secondary Outcome: Percent Change in the Average Daily Pain Score From Baseline to Between Weeks 2 and 12
Description: Percent Change in the Average Daily Pain Score from baseline to between Weeks 2 and 12 measured using Question 5 of the Brief Pain Inventory-Diabetic Neuropathy (BPI-DN). Participants assessed their pain due to diabetes in the last 24 hours on a numeric rating scale from 0 (no pain) to 10 (pain as bad as you can imagine).
Time Frame: Baseline to between Weeks 2 and 12
Population: Intention to Treat (ITT); Baseline Last Observation Carried Forward (BLOCF) imputation was used.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Capsaicin 8% | Placebo
Number analyzed (Participants) | 186 | 183
percentage change | -27.96 (27.25) | -21.00 (29.42)
Statistical Analysis 1: Comparison: Capsaicin 8% vs Placebo; All statistical comparisons were made using two-sided tests at the 5% significance level; Test type: Superiority or Other; p = 0.018, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -7.1, 95% CI 2-sided [-12.9 to -1.2]

3. Secondary Outcome: Weekly Percent Change From Baseline in Average Daily Pain Score
Description: Weekly Percent Change from baseline in average daily pain score from baseline to Week 12 measured using Question 5 of the Brief Pain Inventory-Diabetic Neuropathy (BPI-DN). Participants assessed their pain due to diabetes in the last 24 hours on a numeric rating scale from 0 (no pain) to 10 (pain as bad as you can imagine).
Time Frame: Baseline to Weeks 2, 3, 4, 5, 6, 7, 8, 9,10, 11 and 12
Population: Intention to Treat (ITT ); Baseline last observation carried forward (BLOCF) imputation was used.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Capsaicin 8% | Placebo
Number analyzed (Participants) | 186 | 183
percentage change
  Week 2 | -22.97 (26.24) | -19.00 (27.99)
  Week 3 | -27.17 (27.28) | -20.51 (29.96)
  Week 4 | -28.18 (28.15) | -21.11 (30.52)
  Week 5 | -28.35 (29.48) | -21.17 (30.26)
  Week 6 | -27.87 (30.02) | -21.66 (31.45)
  Week 7 | -29.03 (29.98) | -21.02 (32.50)
  Week 8 | -28.53 (31.92) | -21.46 (31.29)
  Week 9 | -28.61 (31.64) | -21.78 (31.05)
  Week 10 | -28.17 (30.79) | -20.73 (32.39)
  Week 11 | -29.04 (31.13) | -21.75 (32.58)
  Week 12 | -29.64 (31.20) | -20.76 (33.33)
Statistical Analysis 1: Comparison: Capsaicin 8% vs Placebo; Comparison of capsaicin 8% and placebo for change from Baseline to Week 2; Test type: Superiority or Other; p = 0.208, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -4.1, 95% CI 2-sided [-10.4 to 2.3]
Statistical Analysis 2: Comparison: Capsaicin 8% vs Placebo; Comparison of capsaicin 8% and placebo for change from Baseline to Week 3; Test type: Superiority or Other; p = 0.036, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -6.7, 95% CI 2-sided [-13.1 to -0.4]
Statistical Analysis 3: Comparison: Capsaicin 8% vs Placebo; Comparison of capsaicin 8% and placebo for change from Baseline to Week 4; Test type: Superiority or Other; p = 0.027, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -7.2, 95% CI 2-sided [-13.5 to -0.8]
Statistical Analysis 4: Comparison: Capsaicin 8% vs Placebo; Comparison of capsaicin 8% and placebo for change from Baseline to Week 5; Test type: Superiority or Other; p = 0.024, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -7.3, 95% CI 2-sided [-13.6 to -1.0]
Statistical Analysis 5: Comparison: Capsaicin 8% vs Placebo; Comparison of capsaicin 8% and placebo for change from Baseline to Week 6; Test type: Superiority or Other; p = 0.051, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -6.3, 95% CI 2-sided [-12.6 to 0.0]
Statistical Analysis 6: Comparison: Capsaicin 8% vs Placebo; Comparison of capsaicin 8% and placebo for change from Baseline to Week 7; Test type: Superiority or Other; p = 0.012, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -8.1, 95% CI 2-sided [-14.4 to -1.8]
Statistical Analysis 7: Comparison: Capsaicin 8% vs Placebo; Comparison of capsaicin 8% and placebo for change from Baseline to Week 8; Test type: Superiority or Other; p = 0.026, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -7.2, 95% CI 2-sided [-13.5 to -0.8]
Statistical Analysis 8: Comparison: Capsaicin 8% vs Placebo; Comparison of capsaicin 8% and placebo for change from Baseline to Week 9; Test type: Superiority or Other; p = 0.032, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -6.9, 95% CI 2-sided [-13.2 to -0.6]
Statistical Analysis 9: Comparison: Capsaicin 8% vs Placebo; Comparison of capsaicin 8% and placebo for change from Baseline to Week 10; Test type: Superiority or Other; p = 0.020, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -7.5, 95% CI 2-sided [-13.9 to -1.2]
Statistical Analysis 10: Comparison: Capsaicin 8% vs Placebo; Comparison of capsaicin 8% and placebo for change from Baseline to Week 11; Test type: Superiority or Other; p = 0.022, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -7.4, 95% CI 2-sided [-13.7 to -1.1]
Statistical Analysis 11: Comparison: Capsaicin 8% vs Placebo; Comparison of capsaicin 8% and placebo for change from Baseline to Week 12; Test type: Superiority or Other; p = 0.005, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -9.0, 95% CI 2-sided [-15.3 to -2.7]

4. Secondary Outcome: Weekly Average of Average Daily Pain at Baseline and Every Week After Baseline
Description: Weekly average of average daily pain score at Baseline and Weeks 2,4,8 and 12 measured using Question 5 of the Brief Pain Inventory-Diabetic Neuropathy (BPI-DN). Participants assessed their pain due to diabetes in the last 24 hours on a numeric rating scale from 0 (no pain) to 10 (pain as bad as you can imagine).
Time Frame: Baseline and Weeks 2, 4, 8 and 12
Population: Intention to Treat (ITT); Baseline Last Observation Carried Forward (BLOCF) imputation was used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Capsaicin 8% | Placebo
Number analyzed (Participants) | 186 | 183
units on a scale
  Baseline | 6.64 (1.416) | 6.38 (1.473)
  Week 2 | 5.14 (2.059) | 5.14 (2.111)
  Week 4 | 4.83 (2.280) | 5.02 (2.299)
  Week 8 | 4.78 (2.457) | 5.01 (2.343)
  Week 12 | 4.73 (2.436) | 5.08 (2.456)

5. Secondary Outcome: Percentage of Participants With 30% Reduction in Average Daily Pain Score.
Description: Percentage of participants achieving 30% decrease in the average daily pain score in Weeks 2 and 8 and Weeks 2 and 12 measured using Question 5 of the Brief Pain Inventory-Diabetic Neuropathy (BPI-DN). Participants assessed their pain on a numeric rating scale from 0 (no pain) to 10 (pain as bad as you can imagine).
Time Frame: Baseline, Weeks 2-8 and Weeks 2-12
Population: Intention to Treat (ITT ); Baseline last observation carried forward(BLOCF) imputation was used.
Measure: Number; unit: percentage of participants
Arm/Group | Capsaicin 8% | Placebo
Number analyzed (Participants) | 186 | 183
percentage of participants
  30% Pain Reduction-Week 2 to 8 | 74 | 60
  30% Pain Reduction-Week 2 to 12 | 76 | 58
Statistical Analysis 1: Comparison: Capsaicin 8% vs Placebo; Percentage of participants with 30% reduction in average daily pain score assessed in Weeks 2-8. The comparison of the odds ratio of capsaicin 8% to placebo for percent change from baseline was performed using a logistic regression model; Test type: Superiority or Other; p = 0.108, Regression, Logistic; Analysis of regression logistics model including treatment, gender, pain score at baseline, HbA1c at screening and site as factors/covariates; Odds Ratio (OR) = 1.4, 95% CI 2-sided [0.9 to 2.2]
Statistical Analysis 2: Comparison: Capsaicin 8% vs Placebo; Percentage of participants with 30% reduction in average daily pain score assessed in Weeks 2-12. The comparison of the odds ratio of capsaicin 8% to placebo for percent change from baseline was performed using a logistic regression model; Test type: Superiority or Other; p = 0.050, Regression, Logistic; [statistical method as in outcome 5, analysis 1]; Odds Ratio (OR) = 1.5, 95% CI 2-sided [1.0 to 2.4]

6. Secondary Outcome: Percentage of Participants With 50% Reduction in Average Daily Pain Score.
Description: Percentage of participants achieving 50% decrease in the average daily pain score in Weeks 2 and 8 and Weeks 2 and 12 measured using Question 5 of the Brief Pain Inventory-Diabetic Neuropathy (BPI-DN). Participants assessed their pain on a numeric rating scale from 0 (no pain) to 10 (pain as bad as you can imagine).
Time Frame: Baseline, Weeks 2-8 and Weeks 2-12
Population: Intention to Treat (ITT ); Baseline last observation carried forward(BLOCF) imputation was used.
Measure: Number; unit: percentage of participants
Arm/Group | Capsaicin 8% | Placebo
Number analyzed (Participants) | 186 | 183
percentage of participants
  50% Pain Reduction-Week 2 to 8 | 39 | 33
  50% Pain Reduction-Week 2 to 12 | 41 | 35
Statistical Analysis 1: Comparison: Capsaicin 8% vs Placebo; Percentage of participants with 50% reduction in average daily pain score assessed in Weeks 2-8. The comparison of the odds ratio of capsaicin 8% to placebo for percent change from baseline was performed using a logistic regression model; Test type: Superiority or Other; p = 0.403, Regression, Logistic; [statistical method as in outcome 5, analysis 1]; Odds Ratio (OR) = 1.2, 95% CI 2-sided [0.7 to 2.1]
Statistical Analysis 2: Comparison: Capsaicin 8% vs Placebo; Percentage of participants with 50% reduction in average daily pain score assessed in Weeks 2-12. The comparison of the odds ratio of capsaicin 8% to placebo for percent change from baseline was performed using a logistic regression model; Test type: Superiority or Other; p = 0.446, Regression, Logistic; [statistical method as in outcome 5, analysis 1]; Odds Ratio (OR) = 1.2, 95% CI 2-sided [0.7 to 2.0]

7. Secondary Outcome: Overall Participant Status Assessed Using Patient Global Impression of Change (PGIC) Self-assessment Questionnaire in Week 2
Description: Overall participant status assessed using Patient Global Impression of Change (PGIC) self-assessment questionnaire which was used by participants to report on 7 categories listed as follows; Very Much Improved, Much Improved, Minimally Improved, No Change, Minimally Worse, Much Worse and Very Much Worse in Week 2
Time Frame: Baseline to Week 2
Population: Intention to Treat (ITT); Baseline Last Observation Carried Forward (BLOCF) imputation was used.
Measure: Number; unit: participants
Arm/Group | Capsaicin 8% | Placebo
Number analyzed (Participants) | 183 | 180
participants
  Very Much Improved | 10 | 9
  Much Improved | 49 | 38
  Minimally Improved | 72 | 58
  No Change | 45 | 68
  Minimally Worse | 3 | 6
  Much Worse | 3 | 0
  Very Much Worse | 1 | 1
Statistical Analysis 1: Comparison: Capsaicin 8% vs Placebo; Comparing the difference between capsaicin 8% and placebo for counts by category using a Cochran-Mantel-Haenszel test; Test type: Superiority or Other; p = 0.072, Cochran-Mantel-Haenszel; Analysis of Cochran-Mantel-Haenszel test model including treatment, gender, pain score at baseline, HbA1c at screening and site as factors/covariates

8. Secondary Outcome: Overall Participant Status Assessed Using Patient Global Impression of Change (PGIC) Self-assessment Questionnaire in Week 8
Description: Overall participant status assessed using Patient Global Impression of Change (PGIC) self-assessment questionnaire which was used by participants to report on 7 categories listed as follows; Very Much Improved, Much Improved, Minimally Improved, No Change, Minimally Worse, Much Worse and Very Much Worse in Week 8
Time Frame: Baseline to Week 8
Population: Intention to Treat (ITT); Baseline Last Observation Carried Forward (BLOCF) imputation was used.
Measure: Number; unit: participants
Arm/Group | Capsaicin 8% | Placebo
Number analyzed (Participants) | 180 | 172
participants
  Very Much Improved | 20 | 16
  Much Improved | 51 | 36
  Minimally Improved | 58 | 48
  No Change | 47 | 59
  Minimally Worse | 4 | 8
  Much Worse | 0 | 4
  Very Much Worse | 0 | 1
Statistical Analysis 1: Comparison: Capsaicin 8% vs Placebo; Comparing the difference between capsaicin 8% and placebo for counts by category using a Cochran-Mantel-Haenszel test; Test type: Superiority or Other; p = 0.075, Cochran-Mantel-Haenszel; [statistical method as in outcome 7, analysis 1]

9. Secondary Outcome: Overall Participant Status Assessed Using Patient Global Impression of Change (PGIC) Self-assessment Questionnaire in Week 12
Description: Overall participant status assessed using Patient Global Impression of Change (PGIC) self-assessment questionnaire which was used by participants to report on 7 categories listed as follows; Very Much Improved, Much Improved, Minimally Improved, No Change, Minimally Worse, Much Worse and Very Much Worse in Week 12
Time Frame: Baseline to Week 12
Population: Intention to Treat (ITT); Baseline Last Observation Carried Forward (BLOCF) imputation was used.
Measure: Number; unit: participants
Arm/Group | Capsaicin 8% | Placebo
Number analyzed (Participants) | 168 | 172
participants
  Very Much Improved | 23 | 22
  Much Improved | 45 | 29
  Minimally Improved | 39 | 40
  No Change | 50 | 72
  Minimally Worse | 9 | 8
  Much Worse | 2 | 1
  Very Much Worse | 0 | 0
Statistical Analysis 1: Comparison: Capsaicin 8% vs Placebo; Comparing the difference between capsaicin 8% and placebo for counts by category using a Cochran-Mantel-Haenszel test; Test type: Superiority or Other; p = 0.169, Cochran-Mantel-Haenszel; [statistical method as in outcome 7, analysis 1]

10. Secondary Outcome: Change From Baseline in the European Quality Of Life (QOL) Questionnaire in 5 Dimensions (EQ-5D) With Visual Analog Scale (VAS) to Weeks 2, 8 and 12
Description: Change from Baseline in the European Quality Of Life (QOL) questionnaire in 5 dimensions (EQ-5D) with Visual Analog Scale (VAS) to Weeks 2, 8 and 12. EQ-5D self-reported questionnaire is used to measure health-related quality of life by measuring 5 dimensions of health: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The EQ-5D questionnaire includes a visual analog scale (VAS) which records participants self-rated health status on a graduated (0-100) scale with higher scores indicating higher Health-Related Quality of Life (HRQoL).
Time Frame: Baseline to Weeks 2, 8 and 12
Population: Intention to Treat (ITT); Baseline and Last Observation Carried Forward (BLOCF) imputation was used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Capsaicin 8% | Placebo
Number analyzed (Participants) | 186 | 183
units on a scale
  Week 8 [ N=180;N=170] | 4.0 (17.09) | 3.5 (18.36)
  Week 12 [N=170; N=172] | 3.8 (17.94) | 3.7 (19.08)
  Week 2 [N=184; N=181] | 1.3 (15.20) | 3.9 (18.81)
Statistical Analysis 1: Comparison: Capsaicin 8% vs Placebo; The statistical comparison between Baseline and Week 8 was made using two-sided tests at the 5% significance level; Test type: Superiority or Other; p = 0.320, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 1.7, 95% CI 2-sided [-1.6 to 5.0]
Statistical Analysis 2: Comparison: Capsaicin 8% vs Placebo; The statistical comparison between Baseline and Week 12 was made using two-sided tests at the 5% significance level; Test type: Superiority or Other; p = 0.473, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 1.2, 95% CI 2-sided [-2.1 to 4.5]
Statistical Analysis 3: Comparison: Capsaicin 8% vs Placebo; The statistical comparison between Baseline and Week 2 was made using two-sided tests at the 5% significance level; Test type: Superiority or Other; p = 0.514, ANCOVA; LS Mean Difference = 1.7, 95% CI 2-sided [-4.4 to 2.2]

11. Secondary Outcome: Change in Hospital Anxiety and Depression Scale (HADS) Anxiety Scale From Baseline to Weeks 2, 8 and 12
Description: The Hospital Anxiety and Depression Scale (HADS) is a self-report scale developed for the assessment of anxiety and depression, that contain 14 items rated on a 4-point Likert-type scale. There are 2 subscales,one assessing depression and the other anxiety. The 7-item depression and anxiety subscales yield scores of 0 to 21 that are interpreted with the following cut-off points: 0 to 7, normal; 8 to 10, mild mood disturbance; 11 to 14, moderate mood disturbance; and 15 to 21, severe mood disturbance.
Time Frame: Baseline to Weeks 2, 8 and 12
Population: Intention to Treat (ITT); Baseline and Last Observation Carried Forward (BLOCF) imputation was used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Capsaicin 8% | Placebo
Number analyzed (Participants) | 186 | 183
units on a scale
  Week 2 [N=183; N=180] | -0.4 (2.57) | -0.5 (2.74)
  Week 8 [N=178; N=171] | -0.7 (2.72) | -0.6 (3.11)
  Week 12 [N=169; N=169] | -0.9 (2.90) | -0.9 (3.03)
Statistical Analysis 1: Comparison: Capsaicin 8% vs Placebo; Comparing the difference between capsaicin 8% and placebo for change from Baseline at Week 2 was completed using ANCOVA model; Test type: Superiority or Other; p = 0.719, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 0.1, 95% CI 2-sided [-0.5 to 0.7]
Statistical Analysis 2: Comparison: Capsaicin 8% vs Placebo; Comparing the difference between capsaicin 8% and placebo for change from Baseline at Week 8 was completed using ANCOVA model; Test type: Superiority or Other; p = 0.334, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.3, 95% CI 2-sided [-0.8 to 0.3]
Statistical Analysis 3: Comparison: Capsaicin 8% vs Placebo; Comparing the difference between capsaicin 8% and placebo for change from Baseline at Week 12 was completed using ANCOVA model; Test type: Superiority or Other; p = 0.726, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.1, 95% CI 2-sided [-0.7 to 0.5]

12. Secondary Outcome: Change in Hospital Anxiety and Depression Scale (HADS) Depression Scale From Baseline to Weeks 2, 8 and 12.
Description: The Hospital Anxiety and Depression Scale (HADS) is a self-report scale developed for the assessment of anxiety and depression, it contains 14 items rated on a 4-point Likert-type scale. There are 2 subscales,one assessing depression and the other anxiety. The 7-item depression and anxiety subscales yield scores of 0 to 21 that are interpreted with the following cut-off points: 0 to 7, normal; 8 to 10, mild mood disturbance; 11 to 14, moderate mood disturbance; and 15 to 21, severe mood disturbance.
Time Frame: Baseline to Weeks 2, 8 and 12
Population: Intention to Treat (ITT); Baseline and Last Observation Carried Forward (BLOCF) imputation was used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Capsaicin 8% | Placebo
Number analyzed (Participants) | 186 | 183
units on a scale
  Week 2 [ N=184; N=181] | -0.6 (2.39) | -0.6 (2.73)
  Week 8 [N=180; N=171] | -0.7 (2.42) | -0.4 (3.15)
  Week 12 [N=169; N=171] | -0.8 (2.41) | -0.6 (3.24)
Statistical Analysis 1: Comparison: Capsaicin 8% vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p = 0.841, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.1, 95% CI 2-sided [-0.6 to 0.5]
Statistical Analysis 2: Comparison: Capsaicin 8% vs Placebo; [analysis description as in outcome 11, analysis 2]; Test type: Superiority or Other; p = 0.171, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.4, 95% CI 2-sided [-0.9 to 0.2]
Statistical Analysis 3: Comparison: Capsaicin 8% vs Placebo; [analysis description as in outcome 11, analysis 3]; Test type: Superiority or Other; p = 0.595, ANCOVA; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.1, 95% CI 2-sided [-0.7 to 0.4]

13. Secondary Outcome: Treatment Satisfaction Assessment Based on Self-Assessment of Treatment (SAT II) Questionnaire at Baseline, Weeks 8 and 12
Description: Treatment satisfaction assessment based on Self-Assessment Treatment (SAT II) questionnaire and the question "Over the past 7 days, how much has the study treatment improved your pain level?"
Time Frame: Baseline, Weeks 8 and 12
Population: Intention to Treat (ITT); Baseline Last Observation Carried Forward (BLOCF) imputation was used.
Measure: Number; unit: participants
Arm/Group | Capsaicin 8% | Placebo
Number analyzed (Participants) | 186 | 183
participants
  Week 8 [N=177; N=170] [Not at all] | 59 | 82
  Week 8 [N=177; N=170] [Slightly Better] | 35 | 33
  Week 8 [N=177; N=170] [Moderately Better] | 37 | 21
  Week 8 [N=177; N=170] [Quite a Bit Better] | 30 | 21
  Week 8 [N=177; N=170] [Very Much Better] | 16 | 13
  Week 12 [N=166; N=171] [Not at all] | 69 | 91
  Week 12 [N=166; N=171] [Slightly Better] | 30 | 38
  Week 12 [N=166; N=171] [Moderately Better] | 23 | 12
  Week 12 [N=166; N=171] [Quite a Bit Better] | 29 | 14
  Week 12 [N=166; N=171][Very Much Better] | 15 | 16

14. Secondary Outcome: Percent Change in Average Sleep Interference Score From Baseline to Between Weeks 2-8 and Weeks 2-12
Description: Percent change in average sleep interference was measured by Question 9F of the Brief Pain Inventory-Diabetic Neuropathy (BPI DN) and was used to assess pain and sleep interference index. Daily sleep interference rating scale consists of an 11-point numerical scale with which the patient describes how pain related to diabetes has interfered with their sleep during the past 24 hours. On a scale 0 identifies "pain does not interfere with sleep" and 10 identifies "pain completely interferes with sleep". Average sleep interference score is assessed from baseline to Weeks 2-8 and Weeks 2-12.
Time Frame: Baseline, Weeks 2-8 and Weeks 2-12
Population: Intention to Treat (ITT); Baseline Last Observation Carried Forward (BLOCF) imputation was used.
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Capsaicin 8% | Placebo
Number analyzed (Participants) | 186 | 183
percentage of change
  Week 2-8 | -33.12 (33.683) | -24.15 (45.019)
  Week 2-12 | -33.99 (33.566) | -24.67 (43.188)
Statistical Analysis 1: Comparison: Capsaicin 8% vs Placebo; All statistical comparisons were made using two-sided tests at the 5% significance level; Test type: Superiority or Other; p = 0.030, ANCOVA; Analysis of covariance model including treatment,gender, pain score at baseline, HbA1c at screening and site as factors/covariates; LS Mean Difference = -9.0, 95% CI 2-sided [-17.2 to -0.9]
Statistical Analysis 2: Comparison: Capsaicin 8% vs Placebo; All statistical comparisons were made using two-sided tests at the 5% significance level; Test type: Superiority or Other; p = 0.020, ANCOVA; [statistical method as in outcome 14, analysis 1]; LS Mean Difference = -9.5, 95% CI 2-sided [-17.4 to -1.5]

15. Secondary Outcome: Tolerability of Patch Application Assessed by Dermal Assessment on Day 1, 15 Minutes and 60 Minutes After Patch Removal.
Description: Tolerability of patch application was assessed by dermal assessment (0 to 7 point severity score on Dermal Assessment Scale). Data reported is based on the number of participants in the combined category with a score ≥ 4 (Definite edema or higher), 15 and 60 minutes after patch removal.
Time Frame: Day 1, 15 minutes and 60 minutes after patch removal
Population: Safety Analysis Set (SAF)
Measure: Number; unit: participants
Arm/Group | Capsaicin 8% | Placebo
Number analyzed (Participants) | 186 | 183
participants
  15 minutes after patch removal [N=185,N=180] | 0 | 2
  60 minutes after patch removal [N=185,N=179] | 0 | 2

16. Secondary Outcome: Change From Pre-application in"Pain Now" Score
Description: Change from pre-application in"Pain Now" score was measured on a scale from 0-10 where 0 equates to "No Pain" and 10 to "Pain as bad as you can imagine". Participants were asked to provide pain ratings relative only to the area of pain undergoing treatment.
Time Frame: Pre-application and 15 minutes and 60 minutes after patch removal
Population: Safety Analysis Set (SAF)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Capsaicin 8% | Placebo
Number analyzed (Participants) | 186 | 183
units on a scale
  15 minutes after patch removal [N=185; N=183] | -1.6 (2.49) | -2.0 (2.08)
  60 minutes after patch removal [N=185; N=182] | -1.8 (2.57) | -2.2 (2.07)

17. Secondary Outcome: Number of Participants Who Used Rescue Pain Medication Days 1 Through 5
Description: Summarized number of participants who used Rescue Pain Medications for Pain
Time Frame: Days 1 - 5
Population: Safety Analysis Set (SAF)
Measure: Number; unit: participants
Arm/Group | Capsaicin 8% | Placebo
Number analyzed (Participants) | 186 | 183
participants
  Overall | 35 | 10
  Analgesics | 22 | 9
  Anilides | 20 | 9
  Natural opium alkaloids | 14 | 4
  Other opioids | 2 | 0
  Salicylic acid and derivatives | 1 | 0
  Antiinflammatory and antirheumatic products | 15 | 1
  Propionic acid derivatives | 15 | 1
  Other gynecologicals | 15 | 1
  Antiinflammatory products vaginal administration | 15 | 1
  Topical products for joint and muscular pain | 16 | 1
  Antiinflammatory preparations, nonsteroids for top | 15 | 1
  Preparations with salicylic acid derivatives | 1 | 0

18. Secondary Outcome: Safety Assessed Through Adverse Events (AE) and Serious Adverse Events (SAE), Vital Signs, and Laboratory Analyses From Baseline to Week 12
Description: Number of patients assessed for Safety through Adverse Events (AE) and Serious Adverse Events (SAE), vital signs, and laboratory analyses from baseline to week 12
Time Frame: Baseline to Week 12
Population: Safety Analysis Set (SAF)
Measure: Number; unit: participants
Arm/Group | Capsaicin 8% | Placebo
Number analyzed (Participants) | 186 | 183
participants
  Treatment-emergent adverse events (TEAEs) | 87 | 62
  Drug-related TEAEs | 65 | 23
  Deaths | 0 | 0
  Serious TEAEs | 2 | 7
  Drug-related serious TEAEs | 0 | 0
  TEAEs permanent discontinuation of study drug | 0 | 0
  Drug-related TEAEs to permanent discontinuation | 0 | 0
  Application site reactions | 63 | 15

ADVERSE EVENTS:
Time Frame: Adverse Events were reported from the first application of study drug to Week 12 weeks
Arm/Group | Capsaicin 8% | Placebo
Serious Adverse Events (participants affected / at risk) | 2/186 | 7/183
Other Adverse Events (participants affected / at risk) | 61/186 | 18/183
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Capsaicin 8% (N=186) | Placebo (N=183)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Coronary artery disease (Cardiac disorders) | 0 | 1
Noncardiac chest pain (General disorders) | 0 | 1 — Noncardiac chest pain
Postprocedural infection (Infections and infestations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Convulsion (Nervous system disorders) | 1 | 0
Knee arthroplasty (Surgical and medical procedures) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Capsaicin 8% (N=186) | Placebo (N=183)
Application site pain (General disorders) | 18 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 20 | 10
Burning sensation (Nervous system disorders) | 26 | 5

LIMITATIONS AND CAVEATS:
Company makes no warranties or representations of any kind as to the posting, expressed or implied, including warranties of merchantability and fitness for a particular purpose, and shall not be liable for any damages.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish or present trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript at least 30 days prior to publication to ensure that no confidential information of Sponsor is included in the document. Sponsor may delay the publication for an additional 60 days to seek patent protection.